CLINICAL TRIAL: NCT01611896
Title: GRAves Selenium Supplementation Trial (GRASS) - an Investigator-initiated Randomised, Blinded, Multicentre Clinical Trial of Selenium Supplementation Versus Placebo in Patients With Graves' Hyperthyroidism
Brief Title: Selenium Supplementation Versus Placebo in Patients With Graves' Hyperthyroidism
Acronym: GRASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Herlev Hospital (Other); Bispebjerg Hospital (Other); Hvidovre University Hospital (Other); Hillerod Hospital, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Danish Council for Independent Research (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Principal Investigator, Per Cramon, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-4-2012-026; GRASS-DP-240 (Other: Copenhagen Trial Unit); 2007-58-0015, 30-0770 (Other: Danish Data Protection Agency); H-4-2012-026 (Other: Regional Research Ethical Committee for the Capital Region)
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Graves' Hyperthyroidism
Keywords: Graves' hyperthyroidism; Graves' disease; Selenium; Quality of Life; ThyPRO; Autoimmunity
MeSH Terms: conditions — Graves Disease; Autoimmune Diseases | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Active Comparator)
  Interventions: Dietary Supplement: Selenium
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Selenium — 100 µg tablets. The dose of daily supplement of selenium is set at 200 µg (two tablets). The duration of the intervention period is between 24-30 months. This is defined by the time of ATD treatment withdrawal, which is scheduled between approximately 12-18 months after randomisation. Selenium supplementation will continue 12 months after withdrawal of ATD treatment.
  Other Names: 'Selen, organisk selen', produced by Jemo-Pharm A/S
  Arms: Selenium
Other: Placebo — Placebo tablets, identical in regards to size, appearance, taste, smell, and solubility to the experimental intervention tablet will be produced by Jemo-Pharm A/S, http://www.jemo-pharm.dk/frame.cfm/cms/id=977/sprog=2/grp=6/menu=1/ (content as in section: Auxiliary agents). The placebo regimen will be identical to the selenium regimen, but consist of two non-active tablets per day for 24-30 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate if selenium supplementation to the standard treatment with anti-thyroid drugs in patients with Graves' hyperthyroidism, will lead to a fewer people with anti-thyroid treatment failure and faster remission, in terms of better quality of life during the first year of treatment and more patients staying in remission.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Active Graves' hyperthyroidism (suppressed TSH (< 0.1) and positive TRAb) measured within the last two months prior to the inclusion date.
* Written informed consent

Exclusion Criteria:

* Major co-morbidity, making the participants unlikely to continuously receive trial intervention in the intervention period.
* Previous treatment with radioactive iodine.
* Current ATD treatment having been received for more than two months.
* Treatment with immunomodulatory drugs, such as cyclosporine A, methotrexate, cyclophosphamide.
* Allergy towards the components in the selenium and placebo pills.
* Pregnant or breast-feeding women.
* Intake of selenium supplementation above 70 µg per day (70 µg corresponds to the amount in a multivitamin tablet).
* Unable to read and understand Danish.
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with the composite outcome of 'ATD treatment failure' | Last 12 months (± 1 month) of the intervention period
  'ATD treatment failure' is defined as:
  * The participant receives ATD treatment (at any level) during the last 12 months (± 1 month) of the intervention period; or
  * The participant has thyroid hyperfunction (TSH <0.1) during the last 12 months (± 1 month) of the intervention period; or
  * The participant has been referred to ablative therapy (radioactive iodine or thyroid surgery) at some point during the entire intervention period.

SECONDARY OUTCOMES:
Proportion of participants who receives ATD treatment (at any level) during the last 12 months (± 1 month) of the intervention period | Last 12 months (± 1 month) of the intervention period
Proportion of participants who has thyroid hyperfunction (TSH <0.1) during the last 12 months (± 1 month) of the intervention period | Last 12 months (± 1 month) of the intervention period
Proportion of participants who has been referred to ablative therapy (radioactive iodine or thyroid surgery) at some point during the entire intervention period | Intervention period (24-30 months)
Thyroid-specific QoL during the first year after randomisation, and at the end of the intervention period (24-30 months), as measured by the global score in the ThyPRO questionnaire | First year after randomisation, and at the end of the intervention period (24-30 months)
Level of TRAb at 18 months, and at the end of the intervention period (24-30 months) | 18 months, and at the end of the intervention period (24-30 months)
Hyperthyroid symptoms (ThyPRO subscale) during first year after randomisation | First year after randomisation
Eye symptoms (ThyPRO subscale) during first year after randomisation, and at end of the intervention period (24-30 months) | First year after randomisation, and at end of the intervention period (24-30 months)
Number of participants with adverse reactions during the intervention period | Intervention period (24-30 months)
  Participants will be asked to report about known adverse reactions (specified in the protocol) at 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, and 12 months after ATD treatment withdrawal. In addition, participants are instructed to contact their trial contact person in case they experience adverse reactions.
Number of participants with serious adverse events during the intervention period | Intervention period (24-30 months)
  To make sure we get information on serious adverse events, data on hospital admissions and mortality will be obtained through the national databases (the National Patient Registry and the Danish Civil Registration System) at the end of the trial. Also, participants are informed and instructed to contact their trial contact person in case they:
  * are admitted to a hospital for selenium intoxication;
  * experience a clinical picture indicative of selenium intoxication; or
  * experience a clinical picture unexpected, but suspected to be related to selenium intoxication.

CONTACTS AND LOCATIONS:
Overall Officials: Aase K Rasmussen, DMSc, Study Chair — Department of Medical Endocrinology, Rigshospitalet; Torquil Watt, Ph.D., Study Chair — Department of Medical Endocrinology, Rigshospitalet; Laszlo Hegedüs, DMSc, Study Chair — Department of Endocrinology and Metabolism, Odense University Hospital; Steen J Bonnema, Ph.D., Study Chair — Department of Endocrinology and Metabolism, Odense University Hospital; Jeppe Gram, Ph.D., Study Chair — Department of Endocrinology, Hospital of Southwest Denmark; Christian Gluud, DMSc, Study Chair — Copenhagen Trial Unit, Centre for Clinical Intervention Research, Rigshospitalet; Jakob B Bjorner, Ph.D., Study Chair — National Research Centre for the Working Environment, and Institue of Public Health Science, University of Copenhagen; Per Cramon, MD, Principal Investigator — Department of Medical Endocrinology, Rigshospitalet
Locations (8):
- Denmark (8):
  - Department of Endocrinology and Gastroenterology, Bispebjerg Hospital, Copenhagen
  - Department of Medical Endocrinology, Rigshospitalet, Copenhagen
  - Department of Endocrinology, Hospital of Southwest Denmark, Esbjerg
  - Department of Medicine, Gentofte Hospital, Gentofte Municipality
  - Department of Internal Medicine O 106, Endocrine Unit, Herlev Hospital, Herlev
  - Department of Cardiology and Endocrinology, Endocrine Unit, Hillerød Hospital, Hillerød
  - Department of Endocrinology, Section 541, Hvidovre Hospital, Hvidovre
  - Department of Endocrinology and Metabolism, Odense University Hospital, Odense

REFERENCES:
- [Derived] Cramon PK, Winther KH, Boesen VB, Larsen CB, Bjorner JB, Nordqvist SF, Forman JL, Juul AB, Bach-Mortensen P, Knudsen N, Nolsoe RL, Vilsboll T, Andries A, Gram J, Nygaard B, Demircan K, Chillon TS, Schomburg L, Hegedus L, Bonnema SJ, Feldt-Rasmussen U, Rasmussen AK, Watt T. Selenium supplementation in individuals with newly diagnosed Graves' hyperthyroidism: a double-blind, multi-centre RCT. Eur Thyroid J. 2026 Jan 6;15(1):ETJ250264. doi: 10.1530/ETJ-25-0264. Print 2026 Jan 1. PMID 41384622
- [Derived] Cramon P, Rasmussen AK, Bonnema SJ, Bjorner JB, Feldt-Rasmussen U, Groenvold M, Hegedus L, Watt T. Development and implementation of PROgmatic: A clinical trial management system for pragmatic multi-centre trials, optimised for electronic data capture and patient-reported outcomes. Clin Trials. 2014 Jun;11(3):344-354. doi: 10.1177/1740774513517778. PMID 24519964
- [Derived] Watt T, Cramon P, Bjorner JB, Bonnema SJ, Feldt-Rasmussen U, Gluud C, Gram J, Hansen JL, Hegedus L, Knudsen N, Bach-Mortensen P, Nolsoe R, Nygaard B, Pociot F, Skoog M, Winkel P, Rasmussen AK. Selenium supplementation for patients with Graves' hyperthyroidism (the GRASS trial): study protocol for a randomized controlled trial. Trials. 2013 Apr 30;14:119. doi: 10.1186/1745-6215-14-119. PMID 23782950